CLINICAL TRIAL: NCT00894894
Title: Safety Study to Determine the Maximum Tolerated Dose, Pharmacokinetics and Pharmacodynamics of Oral MP470, a Multitargeted Tyrosine Kinase Inhibitor, in Patients With Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGI-0470-01
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumors
Keywords: MP470; MP-470; SuperGen; Tyrosine; Kinase; Inhibitor; Solid Malignancies; Oncology
MeSH Terms: conditions — Neoplasms | interventions — amuvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MP-470 — escalating daily doses of amuvatinib
  Other Names: amuvatinib
Drug: amuvatinib (MP-470) — escalating doses of daily amuvatinib

SUMMARY:
Multicenter, open-label, dose-ranging study in two parts: maximum tolerated dose (MTD) segment (the first 28-day course of MP 470) followed by long-term safety segment.

MTD segment: follows standard oncology phase-I design; within-patient dose level adjustments prohibited; each patient participates in one of three stages:

1. Accelerated Titration Stage
2. Dose Escalation/De-Escalation Stage
3. Dose Confirmation Stage

DETAILED DESCRIPTION:
Multicenter, open-label, dose-ranging study in two parts: MTD Segment (the first 28-day course of MP 470) followed by Long-Term Safety Segment

MTD Segment: follows standard oncology phase-I design; within-patient dose level adjustments prohibited; each patient participates in one of three stages:

Accelerated Titration Stage: 1 patient per dose level; first patient receives MP 470 at 100 mg/day; subsequent patients assigned higher dose levels based on modified Fibonacci sequence; stage stops when any first-course DLT is observed or when grade-2 or greater MP 470-related toxicity is observed at 2 dose levels; dosing next patient prohibited until previous patient's MTD-Segment result is confirmed Dose Escalation/De-Escalation Stage: 3 patients per cohort; two additional patients enrolled to receive last dose level studied during Accelerated Titration Stage (first 3-patient cohort); subsequent 3-patient cohorts assigned dose level conditional on number of patients with first-course DLT in previous cohort; new cohorts enrolled until MTD is defined; dosing next cohort prohibited until previous cohort's MTD-Segment results are confirmed Dose Confirmation Stage: an additional 6-10 patients enrolled to receive MP 470 at the established MTD; patient accrual stops following Dose Confirmation Long-Term Safety Segment: patients continue receiving 28-day courses of MP 470 until experiencing unmanageable toxicity or disease progression; within-patient dose level adjustments based on toxicity; DLT during preceding 28-day course mandates one-level dose reduction; one-level dose increase possible in absence of grade-3 or greater MP 470-related AEs during preceding 28-day course

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a histological or cytological diagnosis of unresectable or metastatic solid-tumor cancer that is refractory to standard therapies or for which no standard therapy exists. Patients with refractory lymphoma (Hodgkin's or NHL) are also permitted to participate.
2. The patient must read, understand and sign the IRB-approved informed consent form (ICF) confirming his or her willingness to participate in this trial.
3. The patient is willing and able to participate in all of the required evaluations and procedures described in this study protocol, including swallowing MP 470 capsules.
4. The patient is at least 18 years old.
5. The patient is capable of fasting for 6 hours.
6. The patient has Karnofsky Performance Status ≥ 70 (see Appendix 5).
7. The patient has adequate bone marrow function evidenced, at minimum, by Hgb ≥ 9 g/dL, ANC ≥ 1.5 x 109/L and platelet count ≥ 100 x 109/L.
8. The patient has normal renal and hepatic function evidenced, at minimum, by total serum bilirubin ≤ 2 mg/dL; AST and ALT ≤ 2.5 x ULN (upper limit of normal for the clinical laboratory), but ≤ 5 x ULN is acceptable if due to hepatic metastases; serum albumin ≥ 2 g/dL; and serum creatinine ≤ 2 mg/dL.
9. The patient has normal cardiac function in the opinion of the investigator and supported by left ventricular ejection fraction (LVEF) 50% or greater on the screening echocardiogram, no significant abnormalities on the screening ECG (eg, left bundle branch block, III degree AV block, acute myocardial infarction or QTc interval > 450 msec) and no history of additional risk factors for torsade de pointes (eg, heart failure, hypokalemia or family history of Long QT Syndrome).
10. The patient has recuperated from any prior surgical procedures including at least 4 weeks rest since a major surgery.
11. The patient does not have childbearing potential or has had a negative serum pregnancy test within the past 14 days.
12. The patient does not have reproductive potential or has agreed to use and will use an approved method of contraception during the study and for 3 months following the last dose of MP 470.
13. The patient is not lactating.

Exclusion Criteria:

1. The patient has a life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of oral MP 470, or put the study outcomes at risk.
2. The patient has any serious, uncontrolled active infection that requires systemic treatment.
3. The patient has a history of significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure and/or myocardial infarction.
4. The patient has received any anticancer agent(s) within the past 3 weeks, including investigational agents, chemotherapy (6 weeks for nitrosoureas or mitomycin), immunotherapy, biologic or hormonal therapy other than LHRH agonists.
5. The patient has received radiation therapy within the past 4 weeks.
6. The patient has a grade-2 or more severe toxicity (other than alopecia) continuing from prior anticancer therapy.
7. The patient has active CNS metastases (primary brain tumors are permitted).
8. The patient requires treatment with immunosuppressive agents other than corticosteroids that have been at stable doses for at least 2 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Translation Genomics Research Institute (TGen)/Scottsdale Clin.Researc, Scottsdale, Arizona
  - So. Texas Accelerated Research Therapeutics-START, San Antonio, Texas

REFERENCES:
- [Derived] Tibes R, Fine G, Choy G, Redkar S, Taverna P, Oganesian A, Sahai A, Azab M, Tolcher AW. A phase I, first-in-human dose-escalation study of amuvatinib, a multi-targeted tyrosine kinase inhibitor, in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2013 Feb;71(2):463-71. doi: 10.1007/s00280-012-2019-3. Epub 2012 Nov 23. PMID 23178951